CLINICAL TRIAL: NCT02263794
Title: Hyperpolarized Magnetic Resonance Imaging in Asthma Pre- and Post-Bronchial Thermoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Grace Parraga (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, University of Western Ontario, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROB0039
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Bronchial Thermoplasty
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Image guided bronchial thermoplasty (Experimental): At pre-treatment Visit 3, imaging data will be acquired to generate a patient-specific bronchial thermoplasty treatment plan which will include 15-20 target airways, prioritized in order of importance and grouped by lobe, to be targeted during a single session BT treatment procedure. Airways demonstrating dynamic or static bronchoconstriction will be targeted for BT treatment based on their spacial proximity to ventilation defects.
  Interventions: Procedure: Image Guided Bronchial Thermoplasty
- Conventional bronchial thermoplasty (Active Comparator): Patients in this group will undergo conventional 3 stage bronchial thermoplasty (during 3 separate bronchoscopies).
  Interventions: Procedure: Conventional Bronchial Thermoplasty

INTERVENTIONS:
Procedure: Conventional Bronchial Thermoplasty — Conventional bronchial thermoplasty is performed during three bronchoscopy sessions each separated by approximately three weeks.
  Arms: Conventional bronchial thermoplasty
Procedure: Image Guided Bronchial Thermoplasty — Patient-specific bronchial thermoplasty based on imaging data will be performed during one bronchoscopy session.
  Arms: Image guided bronchial thermoplasty

SUMMARY:
Patients in London and Hamilton with severe asthma who are deemed eligible by a respirologist to undergo bronchial thermoplasty treatment will be randomized to image-guided or conventional bronchial thermoplasty using hyperpolarized noble gas imaging.

DETAILED DESCRIPTION:
This is a one year, single centre randomized controlled trial. Subjects will be identified through the London Asthma Centre located at St. Joseph's Hospital and from Hamilton at St. Joseph's Healthcare, and will be given a letter of information for the study. The study will only recruit subjects with asthma who are undergoing BT as part of their normal clinical care and asthma treatment plan. Those interested will sign the consent form at the clinic.

Bronchial thermoplasty (BT) is a novel FDA approved outpatient asthma treatment procedure which aims to "cure" symptoms by permanently reducing airway smooth muscle mass in the lobar and segmental bronchi. Under local anesthetic, radiofrequency energy is delivered to warm the airway wall to 65 degrees celcius. The effect of this procedure is a reduction in airway smooth muscle mass in the treated airways resulting in a reduced potential for bronchoconstriction.

Fourteen asthma patients will be enrolled in the study and each subject will visit the centre on five occasions (three pre-treatment visits and two post-treatment visits). We will evaluate pre-therapy optimization using inflammometry, pre-therapy ventilation defect reproducibility and BT treatment effects (pre-treatment visit 1= 5±2 days pre-optimization, pre-treatment visit 2 = 15±7 days pre-BT, pre-treatment visit 3 = 5±2 days pre-BT, post-treatment visit 4=6 weeks post-BT, post treatment visit 5 = 6 months post-BT). At pre-treatment visit 1, patients will be randomized to image-guided or conventional therapy. For all subjects, at all visits, spirometry, plethysmography and 3He and/or 129Xe MRI will be performed. Methacholine challenge (MCh) will be performed (for those subjects with FEV1 >60%) at pre-treatment visit 3 and post-treatment visit 4 with spirometry and MRI performed pre- and post-MCh. Pre-treatment visit 3 will include a low-dose thoracic CT that will be used to generate a detailed 3D model of the airway tree. MRI will be co-registered to the CT with 3D airway rendering to enable spatial comparisons between ventilation defects and airways.

All subjects will also complete bi-weekly and weekly quality of life questionnaires. Self-reported data will be uploaded by each subject monthly to our website using a confidential and password protected upload.

MRI of the lungs will be performed using an inhaled contrast agent: either Hyperpolarized Helium-3 or Hyperpolarized Xenon-129. Participants will inhale the hyperpolarized gas and perform a breathhold for up to 16 seconds. Two different types of images will be acquired in the coronal plain during each visit: 1) 1H thoracic cavity, and 2) 3He and/or 129Xe static ventilation. Respiration and oxygen saturation will be monitored throughout the imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Male and female aged 18-60 years of age with a clinical diagnosis of asthma, as per:

  * Beta-agonist reversibility of FEV1>12%, OR
  * Methacholine FEV1 PC20 ≤ 8 mg/ml if not receiving ICS or ≤ 16mg/ml if receiving an ICS.
* Subject has asthma and is taking regular maintenance medication for the past 12 months that includes:

  * Inhaled corticosteroid (ICS)
  * Long-acting beta agonist (LABA)
  * Other asthma medication such as leukotriene modifier, or anti-IgE, are acceptable
* FEV1 > 50%pred pre-bronchodilator
* Subject assigned by the clinical team to receive bronchial thermoplasty as part of their asthma treatment plan
* Subject is a non-smoker for 1 year or greater (if former smoker less than 10 pack years total smoking history).
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* Subject is judged to be in otherwise stable health on the basis of medical history

Exclusion Criteria:

* Subject is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Subject is unable to perform spirometry or plethysmography maneuvers
* Subject is pregnant
* Recent (within 4 weeks of BL Visit 1) or current asthma exacerbation and/or respiratory tract infection
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.) (At the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Whole lung and lobe specific ventilation defect percent (VDP) as measured by 3He or 129Xe | 48 +/- 2 weeks post bronchial thermoplasty treatment
  Change in VDP post BT

SECONDARY OUTCOMES:
Pulmonary function measurements | 48 +/- 2 weeks post bronchial thermoplasty
  Change in pulmonary function post BT
Quality of Life questionnaires | 48 +/- 2 weeks post bronchial thermoplasty
  Change in subject reported QOL post BT
Dyspnea Scales | 48 +/- 2 weeks post bronchial thermoplasty
  Dyspnea scale score post BT

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario; David G McCormack, MD, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario

REFERENCES:
- [Background] Svenningsen S, Kirby M, Starr D, Coxson HO, Paterson NA, McCormack DG, Parraga G. What are ventilation defects in asthma? Thorax. 2014 Jan;69(1):63-71. doi: 10.1136/thoraxjnl-2013-203711. Epub 2013 Aug 16. PMID 23956019
- [Background] Janssen LJ. Airway smooth muscle as a target in asthma and the beneficial effects of bronchial thermoplasty. J Allergy (Cairo). 2012;2012:593784. doi: 10.1155/2012/593784. Epub 2012 Sep 16. PMID 23024662
- [Background] Pavord ID, Cox G, Thomson NC, Rubin AS, Corris PA, Niven RM, Chung KF, Laviolette M; RISA Trial Study Group. Safety and efficacy of bronchial thermoplasty in symptomatic, severe asthma. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1185-91. doi: 10.1164/rccm.200704-571OC. Epub 2007 Sep 27. PMID 17901415
- [Derived] Capaldi DPI, Guo F, Xing L, Parraga G. Pulmonary Ventilation Maps Generated with Free-breathing Proton MRI and a Deep Convolutional Neural Network. Radiology. 2021 Feb;298(2):427-438. doi: 10.1148/radiol.2020202861. Epub 2020 Dec 8. PMID 33289613
- [Derived] Svenningsen S, Nair P, Guo F, McCormack DG, Parraga G. Is ventilation heterogeneity related to asthma control? Eur Respir J. 2016 Aug;48(2):370-9. doi: 10.1183/13993003.00393-2016. Epub 2016 May 12. PMID 27174885